CLINICAL TRIAL: NCT02525445
Title: Effects of Genuine vs Sham Acupuncture and Communication Type on Relaxation
Acronym: ACU
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Mats Lekander, Professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ACU 2013/80-31
Record Dates: First submitted 2015-08-11; First posted 2015-08-17 (Estimated); Last update posted 2015-08-18 (Estimated); Status verified 2015-08

CONDITIONS: Healthy
Keywords: placebo effects; communication; acupuncture therapy; relaxation
MeSH Terms: conditions — Communication | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- acupuncture positive communication (Active Comparator): Genuine acupuncture needles combined with positive communication regarding the expected treatment effects
  Interventions: Procedure: acupuncture; Procedure: positive communication
- sham acupuncture positive communication (Sham Comparator): Sham acupuncture needles combined with positive communication regarding the expected treatment effects
  Interventions: Procedure: sham acupuncture; Procedure: positive communication
- acupuncture neutral communication (Active Comparator): Genuine acupuncture needles combined with neutral communication regarding the expected treatment effects
  Interventions: Procedure: acupuncture; Procedure: neutral communication
- sham acupuncture neutral communication (Sham Comparator): Sham acupuncture needles combined with neutral communication regarding the expected treatment effects
  Interventions: Procedure: sham acupuncture; Procedure: neutral communication

INTERVENTIONS:
Procedure: acupuncture — acupuncture was administered (sharp needles diameter 0.25 x length 40 mm) bilaterally to the acupuncture point pericardium six (PC6) between the tendons of palmaris longus and flexor carpii radialis at two body-inches (one body-inch approximately 1.5 cm) proximal to the wrist at 0.5 body-inch depth. The therapists manually manipulated the needles three times per treatment by rotating, thrusting or lifting the needles. When the participant reported a sense of numbness or soreness and the therapist noted a minimal muscular contraction around the needle.
  Other Names: invasive acupuncture
  Arms: acupuncture neutral communication; acupuncture positive communication
Procedure: sham acupuncture — sham acupuncture was administrated (blunt needles diameter 0.25 x length 40 mm) bilaterally to a non-acupuncture point four body-inch proximal and one body-inch radial from the PC6 point, with the telescopic non-penetrating Park´s sham needle [20]. Park's credible needle looks identical to a real needle but glides upward into its handle, giving an illusion of penetration. A marking tube, identical for both acupuncture types, held the sham needle in place. The therapists manipulated the needles a few seconds three times per session until the needles touched the skin, but no "needle sensation" occurred, and then lifted the needles up from the skin.
  Other Names: placebo acupuncture
  Arms: sham acupuncture neutral communication; sham acupuncture positive communication
Procedure: positive communication — During the acupuncture treatment the therapist conveyed, at least three out of several positive statements, such as: "Many acupuncture studies have shown excellent results concerning relaxation effects", "Brain imaging studies show that acupuncture treatments affect areas that affect pulse, blood-pressure and muscle tension".
  Arms: acupuncture positive communication; sham acupuncture positive communication
Procedure: neutral communication — During the acupuncture treatment the therapists conveyed, at least three out of several neutral statements, such as: "During treatment you will just lie down and rest and I will not talk so much to you", "We don´t really know if acupuncture is a good method for relaxation effects; thus we need to perform this study",
  Arms: acupuncture neutral communication; sham acupuncture neutral communication

SUMMARY:
The purpose of this study is to investigate if it is possible to influence the participants' expectations to improve outcome, in this particular setting the relaxing effects of one single acupuncture treatment with genuine or sham needles combined with positive or neutral communication regarding expected relaxing effects.

DETAILED DESCRIPTION:
Background It is commonly reported that individuals experience a sense of relaxation during acupuncture treatment. However it is not known if the effects are related to the specific effects of needling or non-specific effects associated with the treatment procedure e.g. the communication with the therapist. It is well known that the way in which patients and clinicians communicate with each other affect treatment outcome, and one of the possible mechanisms to mediate the communication-related treatment outcomes is patient expectations.

Aims The aim of the study is therefore to investigate if it is possible to influence the individuals' expectations to improve outcome; in this particular setting the relaxing effects of one single acupuncture treatment with genuine or sham needles combined with positive or neutral communication regarding expected relaxing effects. The investigators also aim to investigate if different therapists influence how individuals perceive treatment effects, blinding and the communication during treatment with genuine and sham acupuncture.

Procedure Nine therapists performed treatments on voluntary healthy individuals who were randomized to a 30 minute treatment session with a) genuine penetrating acupuncture in traditional acupuncture points or b) non-penetrating sham needles in sham points. Within groups, individuals were further randomized to two communication styles 1) neutral communication or 2) strengthened positive communication regarding expectations concerning relaxing effects.

Outcome measures Perceived degree of expectancy and relaxation was measured directly before and after the treatment. The individuals also rated how they experienced the therapist´s communication style regarding grade of positivity and if they believed that the therapist had given them genuine or sham acupuncture directly after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age
* Able to understand and read/write Swedish

Exclusion Criteria:

* No acupuncture training

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 243 (Actual)
Dates: Start 2013-09; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Change from before treatment to after treatment in subjective report of relaxation (0-100 mm Visual analogue scale) | approximately 5 minutes before treatment and approximately 5 minutes after treatment
  Subjective perception of relaxation measured with a 0-100 mm Visual analogue scale

SECONDARY OUTCOMES:
Change from before treatment to after treatment in subjective report of expectations (0-100 mm Visual analogue scale) | approximately 5 minutes before treatment and approximately 5 minutes after treatment
  Subjective perception of expectation measured with a 0-100 mm Visual analogue scale